CLINICAL TRIAL: NCT03738878
Title: Mechanism(s) Underlying Hypotensive Response to ARB/NEP Inhibition - Aim 1
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: An alternative study was developed to replace this study.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Nancy J. Brown, MD, Ajunct professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB#170762
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Valsartan; sacubitril and valsartan sodium hydrate drug combination; Bradykinin; Substance P; Natriuretic Peptide, Brain; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- valsartan then LCZ696 (Active Comparator): After four-week treatment with valsartan, participants will receive intra-arterial infusions of bradykinin, substance P, and BNP in the presence and absence of sitagliptin.
  Then, after three-week washout and four week therapy with LCZ696, participants will receive intra-arterial infusions of bradykinin, substance P, and BNP in the presence and absence of sitagliptin.
  Interventions: Drug: Valsartan; Drug: LCZ696; Drug: Bradykinin; Drug: Substance P; Drug: BNP; Drug: Sitagliptin
- LCZ696 then valsartan (Active Comparator): After four-week treatment with LCZ696, participants will receive intra-arterial infusions of bradykinin, substance P, and BNP in the presence and absence of sitagliptin.
  Then, after three-week washout and four week therapy with valsartan, participants will receive intra-arterial infusions of bradykinin, substance P, and BNP in the presence and absence of sitagliptin.
  Interventions: Drug: Valsartan; Drug: LCZ696; Drug: Bradykinin; Drug: Substance P; Drug: BNP; Drug: Sitagliptin

INTERVENTIONS:
Drug: Valsartan — oral valsartan
Drug: LCZ696 — oral LCZ696
  Other Names: Entresto
Drug: Bradykinin — Intra-arterial bradykinin at three graded doses
Drug: Substance P — Intra-arterial substance P at three graded doses
Drug: BNP — Intra-arterial BNP at three graded doses
  Other Names: Nesiritide
Drug: Sitagliptin — oral sitagliptin
  Other Names: Januvia

SUMMARY:
The purpose of this study is to test the hypothesis that combined angiotensin receptor blockade (ARB)/neprilysin (NEP) inhibition potentiates the effects of exogenous bradykinin, substance P, and brain natriuretic peptide (BNP) on forearm blood flow or endothelial tissue-type plasminogen activator (t-PA) release compared to ARB alone. A secondary goal is to determine if there is an interactive effect of ARB/NEP inhibition and dipeptidyl peptidase 4 (DPP4) inhibition on responses to these peptides.

DETAILED DESCRIPTION:
After informed consent is obtained, subjects will undergo a screening history and physical exam, and anti-hypertensive medications will be withdrawn. During this period, blood pressure (BP) will be measured every one to three days.

After subjects have been off anti-hypertensive medications for three weeks (four for spironolactone), they will be randomized to four-week treatment with valsartan 160 mg bid (80 mg bid for one week, then 160 mg bid) or LCZ696 200 bid (100 mg bid for one week, then 200 mg bid) in a double-blind fashion. On the morning of the 28th day of study drug, subjects will report to the Vanderbilt Clinical Research Center (CRC) after an overnight fast. Subjects will be studied in the supine position in a temperature-controlled room. They will be instrumented for intra-arterial infusions. Subjects will be given their last dose of study drug. One hour after drug administration, we will measure forearm blood flow (FBF) and give bradykinin, substance P, or BNP. Each peptide will be infused in three graded doses for five minutes. After administration of all three peptides, subjects will be allowed to rest for an hour. Then they will be given a single oral dose of sitagliptin 200 mg and be allowed to rest for 90 minutes. We will repeat baseline measurements and the peptide infusions with an intervening rest period. The four-week study treatment and protocol will be repeated after a three-week washout, until participants complete both arms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with essential hypertension defined as having

   1. untreated, seated systolic blood pressure (SBP) of 130 mmHg or greater on three separate occasions, or
   2. untreated, seated diastolic BP (DBP) of 80 or greater on three separate occasions, or
   3. taken anti-hypertensive agent(s) for a minimum of six months.
2. For female subjects, the following conditions must be met:

   1. postmenopausal status for at least one year, or
   2. status post-surgical sterilization, or
   3. if of childbearing potential, utilization of adequate birth control and willingness to undergo urine beta-human chorionic gonadotropin (hCG) testing prior to drug treatment and on every study day.

Exclusion Criteria:

1. Presence of secondary form of hypertension
2. Symptomatic hypertension and/or SBP>170 mmHg or DBP>110 mmHg, relevant to the washout period
3. History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, angiotensin-converting enzyme inhibitor (ACEi), ARBs, or NEPi, as well as known or suspected contraindications to the study drugs
4. History of angioedema
5. History of pancreatitis or known pancreatic lesions
6. History of significant cardiovascular disease (other than essential hypertension and left ventricular hypertrophy)
7. Symptomatic hypotension and/or a SBP<100 mmHg at screening or <95 mmHg during the study
8. Serum potassium >5.2 mmol/L at screening or >5.4 mmol/L during the study
9. Individuals using oral contraceptives and smokers in order to reduce the risk of thrombosis following arterial line placement
10. History of serious neurologic disease such as cerebral hemorrhage, stroke, seizure, or transient ischemic attack within six months
11. Presence of significant pulmonary disorders
12. Type 1 diabetes
13. Poorly controlled type 2 diabetes mellitus (T2DM), defined as a HgbA1c >9%
14. Hematocrit <35%
15. Impaired renal function [estimated glomerular filtration rate (eGFR) of <30 mL/min/1.73 m2] as determined by the four-variable Modification of Diet in Renal Disease (MDRD) equation, where serum creatinine (Scr) is expressed in mg/dL and age in years: eGFR (mL/min/1.73m2)=175 • Scr-1.154 • age-0.203 • (1.212 if Black) • (0.742 if female)
16. Use of hormone-replacement therapy
17. Breast feeding and pregnancy
18. History or presence of immunological or hematological disorders
19. History of malignancy other than non-melanoma skin cancer
20. Diagnosis of asthma requiring use of inhaled beta agonist more than once a week
21. Clinically significant gastrointestinal impairment that could interfere with drug absorption
22. Impaired hepatic function [aspartate amino transaminase (AST) and/or alanine amino transaminase (ALT) >3.0 x upper limit of normal range]
23. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult, such as arthritis treated with non-steroidal anti-inflammatory drugs
24. Treatment with chronic systemic glucocorticoid therapy within the last year
25. Treatment with lithium salts
26. History of alcohol or drug abuse
27. Treatment with any investigational drug in the one month preceding the study
28. Mental conditions rendering the subject unable to understand the nature, scope, and possible consequences of the study
29. Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of four participants who were enrolled, one was randomized to treatment order and partially completed two study days. One participant met exclusion criteria. Two participants declined to participate after signing the consent form.
Pre-assignment Details: One participant met exclusion criteria. Two participants declined to participate after signing the consent form.
Groups:
- Valsartan Then LCZ696: After four-week treatment with valsartan, participants will receive intra-arterial infusions of bradykinin, substance P, and BNP in the presence and absence of sitagliptin.
  Then, after three-week washout and four-week therapy with LCZ696, participants will receive intra-arterial infusions of bradykinin, substance P, and BNP in the presence and absence of sitagliptin.
  Valsartan: oral valsartan
  LCZ696: oral LCZ696
  Bradykinin: Intra-arterial bradykinin at three graded doses
  Substance P: Intra-arterial substance P at three graded doses
  BNP: Intra-arterial BNP at three graded doses
  Sitagliptin: oral sitagliptin
- LCZ696 Then Valsartan: After four-week treatment with LCZ696, participants will receive intra-arterial infusions of bradykinin, substance P, and BNP in the presence and absence of sitagliptin.
  Then, after three-week washout and four week therapy with valsartan, participants will receive intra-arterial infusions of bradykinin, substance P, and BNP in the presence and absence of sitagliptin.
  Valsartan: oral valsartan
  LCZ696: oral LCZ696
  Bradykinin: Intra-arterial bradykinin at three graded doses
  Substance P: Intra-arterial substance P at three graded doses
  BNP: Intra-arterial BNP at three graded doses
  Sitagliptin: oral sitagliptin
Period: Overall Study
Arm/Group | Valsartan Then LCZ696 | LCZ696 Then Valsartan
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated.
Groups:
- Valsartan Then LCZ696: After four-week treatment with valsartan, participants will receive intra-arterial infusions of bradykinin, substance P, and BNP in the presence and absence of sitagliptin.
  Then, after three-week washout and four week therapy with LCZ696, participants will receive intra-arterial infusions of bradykinin, substance P, and BNP in the presence and absence of sitagliptin.
  Valsartan: oral valsartan
  LCZ696: oral LCZ696
  Bradykinin: Intra-arterial bradykinin at three graded doses
  Substance P: Intra-arterial substance P at three graded doses
  BNP: Intra-arterial BNP at three graded doses
  Sitagliptin: oral sitagliptin
- Total: Total of all reporting groups
Arm/Group | Valsartan Then LCZ696 | LCZ696 Then Valsartan | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] |  | 45 [45 to 45] | 45 [45 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Forearm Blood Flow
Description: Forearm blood flow measured by strain gauge plethysmography before and after intra-arterial peptide infusion
Time Frame: After four-week treatment with each crossover drug
Population: Because the study was terminated data from only one participant are included and no statistical analyses were performed.
Measure: Mean (Full Range); unit: mL/min/100mL
Groups:
- LCZ696: Change in forearm blood flow before and after maximal dose of intraarterial bradykinin during LCZ696.
- Valsartan: Change in forearm blood flow before and after maximal dose of intraarterial bradykinin during valsartan.
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 1 | 1
mL/min/100mL | 2.46 [2.46 to 2.46] | 2.99 [2.99 to 2.99]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the full duration of the study - approximately 12 weeks.
Description: The definition of adverse event and/or serious adverse event does not differ.
Groups:
- LCZ966: Adverse events that occurred on LCZ066 study day
- Valsartan: Adverse events that occurred on valsartan study day.
Arm/Group | LCZ966 | Valsartan
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCZ966 (N=1) | Valsartan (N=1)
hypotension (Vascular disorders) | 1 (1) | 0 (0) — symptomatic decrease in blood pressure below 90 mmHg systolic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT03738878/Prot_SAP_000.pdf